CLINICAL TRIAL: NCT05803772
Title: A Phase II, Randomized, Placebo - Controlled Crossover Proof-of-concept Study to Evaluate Efficacy and Safety of Distal Jejunal-release Dextrose Beads Formulation (APHD-012) in Subjects With a Pathological Oral Glucose Tolerance Test (OGTT)
Brief Title: A Study to Evaluate Efficacy and Safety of Distal Jejunal-release Dextrose Beads Formulation in Subjects With a Pathological Oral Glucose Tolerance Test
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aphaia Pharma US LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAP2022-1
Record Dates: First submitted 2023-03-24; First posted 2023-04-07 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: PreDiabetes; Glucose Tolerance Impaired
Keywords: OGTT; Glucose Tolerance; Prediabetes
MeSH Terms: conditions — Prediabetic State; Glucose Intolerance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active to Placebo Cross (Other): Participants will first receive a single dose of APHD-012 12 g daily, under fasting conditions prior to main daily meals for 6 weeks (day 1-42), followed by washout period of 4 weeks (day 43-70), and subsequent crossover to the other treatment APH-012P for 6 weeks (day 71-112).
  Interventions: Drug: APHD-012; Drug: APH-012P
- Placebo to Active Cross (Other): Participants will first receive a single dose of APH-012P daily, under fasting conditions prior to main daily meals for 6 weeks (day 1-42), followed by washout period of 4 weeks (day 43-70), and subsequent crossover to the other treatment APHD-012 12 g for 6 weeks (day 71-112).
  Interventions: Drug: APHD-012; Drug: APH-012P

INTERVENTIONS:
Drug: APHD-012 — Drug: APHD-012 Distal jejunal-release dextrose beads (Aphaia technology, AT)
  Other Names: Distal jejunal-release dextrose beads
Drug: APH-012P — Distal jejunal-release placebo beads
  Other Names: Placebo

SUMMARY:
The primary purpose of the study is to evaluate the efficacy and safety of APHD-012 (distal jejunal-release dextrose [Aphaia technology, AT]) in participants with pre-diabetes (pathological Oral Glucose Tolerance Test (OGTT)).

DETAILED DESCRIPTION:
The goal of this Phase II, Randomized, Placebo-Controlled Crossover Proof-of-Concept Study is to evaluate the efficacy of APHD-012 in patients with pre-diabetes (pathological Oral Glucose Tolerance Test (OGTT)). The main questions it aims to answer are:

1. Are there changes in baseline in Area Under the Curve from Time 0 to 2 Hours (AUC0-2) values of Oral Glucose Tolerance Test (OGTT)?
2. Are there changes in biomarkers (e.g. fasting plasma glucose, Homeostatic Model Assessment for Insulin Resistance (HOMA-IR))?

Participants will receive study medication or placebo once daily for 6 weeks, followed by washout period of 4 weeks, and subsequent crossover to the other treatment arm for 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects 18 - 70 years of age
* Fully vaccinated against SARS-CoV-2.
* Body mass index 25-35 kg/m2
* Subjects with an impaired glucose tolerance defined as: HbA1c values ≥5.7% and ≤ 6.4%, and/or, Impaired glucose tolerance (glucose between 140 and 199 mg/dL at the 2 hours of the Oral Glucose Tolerance Test (OGTT)) with or without impaired fasting glucose (fasting glucose between 100 and 125 mg/dL)
* Stable body weight: gain or loss in body weight ≤ 5% body weight over last 3 months
* History of at least one unsuccessful effort of lifestyle modification to loose >5% of body weight, completed at least 3 months prior to screening. Subject may have been treated with either diet or exercise alone.
* Willingness to undergo screening and all study procedures and examinations (i.e., physical examinations and laboratory investigations before and after the treatment periods) and to wear a flash glucose monitoring device.
* Ability to comprehend subject information and willingness to sign the informed consent.

Exclusion Criteria:

* Evidence of type 2 diabetes defined by fasting plasma glucose ≥ 126 mg/dL; 2-hour OGTT glucose ≥ 200 mg/dL
* Type I diabetes mellitus
* HbA1c ≥ 6.5%
* History of proliferative retinopathy or maculopathy
* Active COVID-19 infection proven by antigen positive Covid Test
* Treatment with any medication for weight loss within the past 3 months before screening.
* Prior or planned weight loss surgery for obesity
* Recent (within past 12 months) or planned endoscopic treatment for obesity.
* Proven history of bulimia or anorexia nervosa
* Eating habits consisting of eating relevant amounts of food throughout the night (after 10 p.m.; except if working on night shifts)
* Treatment with injectable anti-diabetic medications in the last 3 months (e.g., GLP-1 receptor agonists, insulin)
* Treatment with dipeptidyl peptidase-4 inhibitors in the last 3 months
* Confirmed medical history of liver cirrhosis
* Positive test on Viral hepatitis (HbsAG, HCV)
* Positive test on Human immunodeficiency virus (HIV)
* Cholestatic disease
* Alcohol-related liver disease including alcoholic fatty liver, alcoholic hepatitis and alcoholic cirrhosis evidenced by confirmed history of alcohol use, abnormal liver function tests defined below, and complete blood count (CBC), and/or liver biopsy.
* Abnormal liver function tests:

  * Transaminases: Alanine aminotransferase (ALT) ≥ 3x upper limit of normal (ULN); or Aspartate aminotransferase (AST) ≥ 3x ULN;
  * or Alkaline phosphatase (ALK) ≥2.5 x ULN
  * or Total bilirubin ≥2 x ULN
* Stage 4 hypertension (systolic blood pressure (SBP) ≥ 180, diastolic BP (DBP) ≥ 110)
* History or presence of any uncontrolled cardiovascular, pulmonary, hepatobiliary, renal, hematological, gastrointestinal, endocrinologic, immunologic, dermatologic, neurological, psychiatric, metabolic, musculoskeletal, or malignant disease (except conditions accepted for inclusion) which the clinical investigator considers a disqualification for participation in the study.
* Prior or current treatment with drugs aimed to treat abnormal glucose homeostasis including oral antidiabetics, incretin analogues and/or insulin.
* History of uncontrolled illness (e.g. depression, psychosis) or behaviour that at the discretion of the investigator might confound the study results or pose additional risk in administering the study procedures.
* Illicit drug abuse
* Alcohol abuse
* Participation in another investigational drug/biologic or medical device study within 30 days of screening or will be enrolled in another investigational drug or medical device study or any study in which active subject participation is required outside normal hospital data collection during the course of the study.
* Failure to provide informed consent.
* Unwillingness or inability to comply with the study protocol or study-related procedures.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2023-03-31 (Actual); Primary Completion 2024-02-12 (Actual); Study Completion 2024-02-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in AUC0-2h values of Oral Glucose Tolerance Test (OGTT) as measured in blood samples | Day 1 to Day 42; Day 71 to Day 112
  The primary efficacy endpoint is the change from baseline in AUC0-2h values of Oral Glucose Tolerance Test (OGTT) measured in blood samples at the end of each study period (Day 42 and Day 112, respectively). Two baselines will be defined for each period separately (Day 1 and Day 71, respectively).

SECONDARY OUTCOMES:
Change from baseline in fasting plasma glucose concentrations | Day 1 to Day 42; Day 71 to Day 112
  Change from baseline in fasting plasma glucose concentrations will be measured as ratio to baseline of fasting plasma glucose concentration at week 6 of each study period.
Change from baseline in HOMA IR | Day 1 to Day 42; Day 71 to Day 112
  Change from baseline in HOMA IR will be measured as ratio to baseline of HOMA-IR at week 6 of each study period
Number of Participants Reported with At least One Treatment Emergent Adverse Event (TEAE) | Day 1 to Day 42; Day 71 to Day 112
  A treatment-emergent adverse event is defined as any event not present prior to the initiation of the drug treatment or any event already present that worsens in either intensity or frequency following exposure to the drug treatment

OTHER OUTCOMES:
Change in systolic blood pressure (SBP) | Day 1 to Day 42; Day 71 to Day 112
Change from baseline in Diastolic blood pressure (DBP) | Day 1 to Day 42; Day 71 to Day 112
Change from baseline in Heart rate (HR) | Day 1 to Day 42; Day 71 to Day 112
Change from baseline in Triglycerides | Day 1 to Day 42; Day 71 to Day 112
Change from baseline in Cholesterol (Total, LDL, HDL) | Day 1 to Day 42; Day 71 to Day 112
Change from baseline in Fasting plasma insulin | Day 1 to Day 42; Day 71 to Day 112
Change from baseline in HbA1c | Day 1 to Day 42; Day 71 to Day 112
Change from baseline in Alanine transaminase (ALT) | Day 1 to Day 42; Day 71 to Day 112
Change from baseline in Aspartate transaminase (AST) | Day 1 to Day 42; Day 71 to Day 112
Change from baseline in Gamma Glutamyl Transferase (GGT) | Day 1 to Day 42; Day 71 to Day 112
Change from baseline Daily average glucose as measured by Flash Glucose Monitoring (FGM) | Day 1 to Day 42; Day 71 to Day 112
Change from baseline in AUC0-2h of OGTT as measured by Flash Glucose Monitoring (FGM) | Day 1 to Day 42; Day 71 to Day 112

CONTACTS AND LOCATIONS:
Locations (3):
- Slovakia (3):
  - Cell-B s.r.o., Levice, Slovenska
  - ALIAN, s.r.o., Bardejov
  - MEDISPEKTRUM s.r.o., Bratislava

IPD SHARING:
Plan to Share IPD: No